CLINICAL TRIAL: NCT05572190
Title: A Phase 1, Randomized, Open-Label, 2-Part Study to Evaluate the Safety and Pharmacokinetics of ETR028 Acetate and ETR029 Acetate in Healthy Adult Subjects
Brief Title: Evaluate the Safety and Pharmacokinetic Profile of ETR028 and ETR029 in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elysium Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry); Charles River Laboratories International Inc. (Unknown); National Institute on Drug Abuse (NIDA) (NIH); Ohio Third Frontier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: O2P-001; R01DA046102 (NIH)
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- A1.1. 30 mg ETR028 Sentinel (Experimental): 30 mg ETR028 single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A1.1. 30 mg ETR029 Sentinel (Experimental): 30 mg ETR029 single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A1.1. 5 mg HCBT (Active Comparator): 5 mg hydrocodone bitartrate (HCBT) single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A1.1. 10 mg HCBT (Active Comparator): 10 mg HCBT single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A1.2. 30 mg ETR028 (Experimental): 30 mg ETR028 single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A1.2. 30 mg ETR029 (Experimental): 30 mg ETR029 single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A2. <=60mg ETR028 (Experimental): <=60 mg ETR028 single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- A2. <= 80mg HCBT (Active Comparator): <= 80mg HCBT single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B1. [ETR028 + ETR029] blend "1" (Experimental): [ETR028 - dose To Be Determined (TBD) + ETR029 - <=30mg] single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B1. [ETR028 + ETR029] blend "2" (Experimental): [ETR028 - dose TBD + ETR029 - <=30mg] single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B2. [ETR028 + ETR029] blend "3" (Experimental): [ETR028 - dose TBD + ETR029 - <=30mg] single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B2. [ETR028 + ETR029] blend "4" (Experimental): [ETR028 - dose TBD + ETR029 - <=30mg] single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B3. [ETR028 + ETR029] blend "1", "2", "3", or "4" (fed) (Experimental): [ETR028 - dose TBD + ETR029 - <=30mg] single oral dose (fed)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B3. [ETR028 + ETR029] blend "1", "2", "3", or "4" (fasted) (Experimental): 2-fold higher dose of [ETR028 + ETR029] blend "1", "2", "3", or "4" single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B4. [ETR028 + ETR029] blend "1", "2", "3", or "4" (Experimental): 4-fold higher dose of [ETR028 + ETR029] blend "1", "2", "3", or "4" single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B5. [ETR028 + ETR029] blend "1", "2", "3", or "4" (Experimental): 8-fold higher dose of [ETR028 + ETR029] blend "1", "2", "3", or "4" single oral dose (fasted)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT
- B6. [ETR028 + ETR029] blend "1", "2", "3", or "4" (Experimental): 8-fold higher dose of [ETR028 + ETR029] blend "1", "2", "3", or "4" single oral dose (fed)
  Interventions: Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT

INTERVENTIONS:
Drug: ETR028, ETR029, [ETR028 + ETR029] or HCBT — Hydrocodone prodrugs
  Other Names: O2P hydrocodone

SUMMARY:
The goal of this Phase 1 clinical study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of O2P (Oral Overdose Protected) hydrocodone prodrugs (ETR028 and ETR029) relative to hydrocodone bitartrate hemipentahydrate (HCBT) comparator following single oral doses in healthy adult subjects under fasted and fed conditions with naltrexone blockade

DETAILED DESCRIPTION:
This is a Phase 1, randomized, single-site, open-label, single dose, 2-part study to evaluate the safety and PK of immediate release O2P hydrocodone (comprised of prodrug ETR028 or a blend of ETR028 and ETR029 prodrugs) against an HCBT comparator in healthy adult subjects when administered under fasted and fed conditions with naltrexone blockade. Up to approximately 78 healthy adult subjects are planned to be enrolled with each subject participating in 1 treatment period except for subjects in O2P hydrocodone treatment periods crossed over to receive O2P hydrocodone under fed conditions.

ELIGIBILITY:
Inclusion Criteria: Subjects who meet all of the following criteria will be eligible to participate in the study:

1. Subjects must be male or female, 18 to 55 years of age, inclusive, at the Screening Visit;
2. Subjects must be willing and able to give written informed consent for participation in the study prior to the initiation of any screening or study-specific procedures;
3. Subjects must have a body mass index (BMI) within the range of 18 kg/m2 to 32 kg/m2(> 45 kg), inclusive;
4. Subjects must be in general good health, based upon the results of medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG), as judged by the Investigator;
5. Subjects must have an estimated glomerular filtration rate (eGFR) of >= 60 mL/min/1.73 m2 at the Screening Visit. One retest of the exclusionary eGFR value is allowed at the discretion of the Investigator;
6. Subjects must have normal hematologic function at the Screening Visit, defined as the following:

   o Hemoglobin >= 11.5 (female) or >= 12.5 (male); Note: Subjects with non-clinically significant out-of-range values may be rescreened once for purposes of determining study eligibility.
7. Subjects must have all safety laboratory parameters (serum chemistry, hematology, and urinalysis) within normal limits (laboratory reference range) at the Screening and Check-in (Day -1) Visit or, if outside of the normal limits, must meet both of the following criteria:

   * Considered by the Investigator to not be clinically significant; and
   * Abnormal liver function test results (alanine aminotransferase, aspartate aminotransferase, or total bilirubin level) must be < 1.5 × upper limit of normal of the laboratory reference range.

   Note: Subjects with non-clinically significant out-of-range values may be rescreened once for purposes of determining study eligibility.
8. Subjects must confirm they have previously tolerated prescription opioids;
9. Female subjects of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, bilateral salpingectomy, and/or bilateral oophorectomy at least 26 weeks prior to the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone (FSH) in the postmenopausal range at the Screening Visit based on the central laboratory's ranges;
10. Female subjects of childbearing potential must not be pregnant, lactating, or planning a pregnancy from the Screening Visit to 30 days after administration of the last dose of study drug and must have a negative serum pregnancy test result at the Screening Visit and a negative urine pregnancy test result at Day -1 of each treatment period;
11. Female subjects of childbearing potential (i.e., ovulating, premenopausal, and not surgically sterile) with male partners must agree to use a medically accepted contraceptive regimen during their participation in the study and for 30 days after the last administration of study drug. All male subjects with female partners of childbearing potential must agree to use a medically accepted contraceptive regimen during their participation in the study and for 90 days after the last administration of study drug. Medically accepted contraceptive methods are defined as those with 90% or greater efficacy;

    * For male subjects enrolled in the study:

      * Condoms with spermicide; or
      * Surgical sterilization (vasectomy) of the subject at least 26 weeks prior to the Screening Visit.
    * For female subjects enrolled in the study:

      * Intrauterine device for at least 12 weeks prior to the Screening Visit;
      * Hormonal contraception (oral, implant, injection, ring, or patch) for at least 12 weeks prior to the Screening Visit;
      * Diaphragm used in combination with spermicide; or
      * Male partner using condom with spermicide.
12. Male subjects must agree to abstain from sperm donation during the study and through 90 days after administration of the last dose of study drug;
13. Subjects must be willing and able to consume the entire high-fat standardized meal in the designated timeframe required in Parts A and B; and
14. Subjects must be willing to comply with all study procedures and requirements throughout the duration of the study.

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Subjects with a history or presence of significant cardiovascular, hepatic, renal, hematologic, gastrointestinal, infectious, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, or have any other condition that in the opinion of the Investigator, could potentially impact the safety of the subject or metabolism of the study drug;
2. Subjects with a clinically significant history or presence of any gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), liver or kidney disease, gastric bypass, gastric stapling, use of Lapband, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug;
3. Subjects who are positive for hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV), or hepatitis C virus antibody (HCVAb) at the Screening Visit;
4. Subjects who have a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day) within 2 years prior to the Screening Visit or are unwilling to agree to abstain from alcohol and drugs throughout the study;
5. Subjects with positive screen results for drugs of abuse, alcohol, or cotinine at Screening or Check-in (Day -1) Visit;
6. Subjects who have lost or donated > 480 mL of whole blood or blood products within 60 days prior to the Screening Visit;
7. Subjects who have used any prescription or over-the-counter medication or vitamins/herbal supplements (with the exception of hormonal contraceptives and sporadic use of acetaminophen or ibuprofen) within 7 days or 5 half-lives (whichever is longer) prior to randomization until completion of the End of Study Visit, and that in the Investigator's opinion may impact subject safety or the validity of the study results; Note: Within 14 days if the drug is known or suspected to effect hepatic or renal clearance capacity or if the drug is known to be a potential moderate or strong inhibitor/inducer of cytochrome P450 enzymes (e.g., barbiturates, phenothiazine, cimetidine, carbamazepine, etc).18 Vaccinations, including the Coronavirus Disease of 2019 (COVID-19) vaccine, are allowed as long as the vaccines are administered at least 72 hours prior to Check-in (Day -1) Visit.
8. Subjects who have used medications that affect gastrointestinal motility, gastric emptying, or gastric pH (potential hydrogen), such as metoclopramide, proton pump inhibitors, and/or H2 blockers, within 14 days prior to randomization until completion of the End of Study Visit;
9. Subjects who have used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, chewing tobacco, nicotine patch, or nicotine gum) within 28 days prior to Check-in (Day -1) Visit;
10. Subjects who have a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Check-in (Day -1) Visit;
11. Subjects who have clinically relevant abnormal physical findings, ECG, or laboratory values at or during the Screening Visit that, in the opinion of the Investigator, could interfere with the objectives of the study or the safety of the subjects;
12. Subjects with a known hypersensitivity to any component in the formulations of hydrocodone or other opioids;
13. Subjects with any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subjects' participation in the study;
14. Subjects must not consume beverages and foods containing alcohol, poppy seeds, or caffeine/xanthine, or energy drinks from 24 hours prior to Check-in (Day -1) Visit until after the last sample collection of each treatment period;
15. Subjects must not consume products containing grapefruit from 48 hours prior to Check-in (Day -1) Visit until after the last sample collection of each treatment period;
16. Subjects must not engage in strenuous exercise from 48 hours prior to Check-in (Day -1) Visit until after the last sample collection of each treatment period; or
17. Subjects who have used any other investigational product or participated in another research study within a period of 5 half-lives of the product, or a minimum of 30 days prior to study drug administration (whichever is longer).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile | Time Zero (just prior to dose) to 48 hours post dose Timepoints: pre-dose and at 0.5,1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose.
  Plasma concentration-time profile (ng/ml) of ETR028, ETR029, [ETR028 + ETR029] blend, O2P hydrocodone-derived 3 major metabolites (e.g., 3-hydroxy-arylguanadine [3-HAG], 4-hydroxy-arylguanadine [4-HAG], and ETR106), and hydrocodone
Subjects reporting at least one Adverse Event (AE) | From the time a subject is dosed until 8 day post-dose Follow-Up Visit
  An AE can be any unfavorable and/or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the investigational medicinal product, whether or not related to the investigational medicinal product.
Subjects reporting at least one Serious Adverse Event (SAE) | From the time a subject is dosed up to 30 days post-dose
  A Serious Adverse Event is an AE that results in any of the following outcomes; Death, Life-threatening, inpatient hospitalization or causes prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, important medical event (i.e., based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent 1 of the outcomes listed above)

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace, Inc.; Lynn Webster, MD, Study Director — Elysium Therapeutics, Inc.
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No